CLINICAL TRIAL: NCT03122015
Title: The Use of Therapeutic Clown in Painful Procedures in Children: A Pilot Study
Brief Title: The Use of Therapeutic Clown in Painful Procedures in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: St. Justine's Hospital (Other)
Responsible Party: Principal Investigator, Patricia Laforce, Registered nurse, Master's degree student, St. Justine's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-1398
Record Dates: First submitted 2017-04-10; First posted 2017-04-20 (Actual); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Pain, Acute
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Intervention Model Description: This pilot study will include a group that will receive the intervention of distraction by the therapeutic clown (CT) and the other that will receive the standard treatment. The study will take place at St. Justine's Hospital, precisely at the infectious diseases clinic. Recruitment of participants will be by convenience from parents and children who will be eligible for study. The sample of this pilot project will contain approximately 24 children in addition to parents and the nurse who will perform the painful procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Therapeutic clown distraction (Experimental): The child will interact with the therapeutic clown throughout the painful procedure. The types of distraction interventions will be determined by the clown according to the child's age, culture and behavior. The clown can use different distraction activities such as magic, humor, visualization and play. According to various writings, the presence of the clown before the procedure varied between two to 20 minutes. In our study, the presence of the clown with parents and children will be about 10 minutes before the procedure and while the nurse performs the procedure until the child leaves the room. The distraction performed by a therapeutic clown is used in St. Justine' Hospital. Indeed, a team of therapeutic clowns is present in the hospital four times a week to distract the children. However, this procedure is not applied routinely in painful procedures and no study has evaluated its usefulness or effect.
  Interventions: Other: Therapeutic clown distraction
- Standard care (No Intervention)

INTERVENTIONS:
Other: Therapeutic clown distraction — The presence of the therapeutic clown, which can adapt his interventions of distraction to the state of health of the patient and the culture of the child, is a multimodal and multi sensorial distraction intervention and can have an impact on health status, procedures, family and multidisciplinary team members. The results of five studies evaluated the effects of distraction by the clown therapy demonstrate a decrease in pain and anxiety in children aged 2 to 17 years, as well as parental anxiety in painful procedures involving needles such as venipuncture.
  Arms: Therapeutic clown distraction

SUMMARY:
Children in hospitals are frequently subjected to painful procedures, including those involving needles, which are a common source of pain in children. In addition, procedural pain and anxiety can lead to various consequences for the child, as well for the parent and the nurse performing the procedure. The use of physical and psychological interventions is recommended for optimal relief of procedural pain. Moreover, these interventions can be used alone or in combination with pharmacological treatment. Although several analgesics exist and are used in clinical practice, nonpharmacological interventions aimed at the psychological component of pain are not well known and are not always used by the nurses in the pediatric practice. Distracting interventions are widely studied in the literature as it is an effective psychological intervention in the relief of pain and anxiety in children during needle-related pain procedures. The distraction by the therapeutic clown is a multi-modal intervention with multi-sensory effects and appears promising in pain relief and procedural anxiety, but not much studies have been done in the context above. The therapeutic clown can adapt to the age of the child, its culture, its reality of care and can prepare the child for painful procedures. The aim of this study is to assess the feasibility, acceptability and preliminary effects of distraction by therapeutic clown on pain and anxiety of children aged two to 17 years and the level of anxiety of the parents and nurses during a painful procedure in children.

OBJECTIFS AND QUESTIONS:

1. Assess the feasibility and acceptability of distraction by therapeutic clown with children during painful procedures. a) Is the distraction intervention by the therapeutic clown feasible and acceptable during painful procedures?
2. Assess the preliminary effects of distraction by therapeutic clown on pain and anxiety of children and the anxiety of parents and nurses. a) What are the preliminary effects of the therapy clown distraction on children's pain and anxiety, and the anxiety of parents and nurse.

DETAILED DESCRIPTION:
1. BACKGROUND

   1.1 Hospitalized children under 18 years old are frequently undergo painful procedures including needles. Although children often have interventions to relieve pain during the period of hospitalization, few interventions are implemented specifically for painful procedures. Studies show that pain and anxiety associated with the painful procedure, such as needles, can lead to various physiological, physical and psychological consequences in children, as avoidance of medical care. In addition, physiological and psychological effects such as increased heart rate, blood pressure, and anxiety levels were also noted with parents who accompanied their child during a painful procedure. These effects on parents increase the anxiety of the child, which amplifies the pain felt by the child.

   Moreover, the effects of procedural pain do not only affect the child and his parents. Studies reveal that these painful procedures result in impotence and an increased level of anxiety among professionals performing the procedures, which in turn have an impact on children's anxiety and pain. Finally, procedural pain can lead to a lack of collaboration between the child, increasing the length of the procedure and the need for staff.

   1.2 A Canadian study found that pharmacological interventions are widely used among hospitalized children who are experiencing painful procedures but very few non-pharmacological interventions are were used. However, since pain is a multi-sensory experience and emotional and cognitive components modulate nociceptive treatment, the use of analgesics alone cannot alleviate each of the components of pain. Therefore, the use of physical and psychological interventions is recommended for optimal relief of procedural pain. Moreover, these interventions can be used alone or in combination with pharmacological treatment.

   1.3 Among non-pharmacological interventions, distraction interventions are widely studied and recommended for pain and anxiety management experienced in children and adolescents during needle-related pain procedures. Therapeutic clown distraction is a form of distraction, as it has multi-sensory effects that appear promising in children's procedural pain and anxiety management but have been little studied in this context.

   1.4 The presence of the therapeutic clown, which can adapt his interventions of distraction to the state of health of the patient and the culture of the child, is a multimodal and multi sensorial distraction intervention and can have an impact on health status, procedures, family and multidisciplinary team members. The results of five studies evaluated the effects of distraction by the clown therapy demonstrate a decrease in pain and anxiety in children aged 2 to 17 years, as well as parental anxiety in painful procedures involving needles such as venipuncture.
2. AIM The aim of this study is to assess the feasibility, acceptability and preliminary effects of distraction by therapeutic clown on pain and anxiety of children aged 7 to 17 years, and the anxiety of parents and nurses during a painful procedure in children.

OBJECTIFS AND QUESTIONS:

1. Assess the feasibility and acceptability of distraction by therapeutic with children during painful procedures. a) Is the distraction intervention by the therapeutic clown feasible and acceptable during painful procedures?
2. Assess the preliminary effects of distraction by therapeutic clown on the pain and anxiety of children and the anxiety of parents and nurses.

   1. What are the preliminary effects of the therapy clown distraction on children's pain and anxiety, and the anxiety of parents and nurses?

      HYPOTHESES

   <!-- -->

   1. Therapeutic clown distraction is a feasible and acceptable method for procedural pain relief of children.

      3. METHODS

      4.1 Design.

      Experimental before and after pilot study.

      4.2 Sample and Setting.

      This pilot study will include a group that will receive the intervention of distraction by the therapeutic clown (CT) and the other that will receive the standard treatment. The study will take place at St. Justine's Hospital, precisely at the infectious diseases clinic. Recruitment of participants will be by convenience from parents and children who will be eligible for study. The sample of this pilot project will contain approximately 24 children in addition to parents and the nurse who will perform the painful procedure.

      4.3. Measures. Measures of anxiety will be recorded at T1, T2 and general anxiety will be asses by parents after the procedure at T3. Measures for procedural pain will be taken at: T2, during the procedure. Acceptability will be assessed with parents and nurses using an satisfaction survey at T3, after the procedure.

      4.4 Data analysis plan. The characteristics of children, parents and nurses will be described using descriptive statistics. Inferential nonparametric statistics will be used to compare the data of each group and to evaluate the preliminary effects of interventions on child pain and anxiety and parental and nurse anxiety.

      FEASIBILITY

      Acceptability will be assessed with parents and nurses using an satisfaction survey. The questionnaire will be provided to parents in paper form and will be verbally completed by the nurse. In addition, to document the feasibility and acceptability of the study, the number of children participating, as well as the duration of the procedure and the number of professionals involved will be noted throughout the procedure. In the case where the child must receive several vaccines, only the first immunization will be timed.

      4. POSSIBLE PITFALLS AND SOLUTIONS

      Since this study represents a pilot study, the results cannot be generalized and will not allow us to determine whether one intervention will be more effective than the other.

      5. CONTRIBUTION AND EXPECTED RESULTS

      These interventions, which we believe are feasible, could help reduce the negative impact of painful procedures on children, parents and nurses.

ELIGIBILITY:
Inclusion Criteria:

* Children requiring immunization.
* Understand and speak French or who are accompanied by someone who understands and speaks french.
* Children accompanied by at least one parent.

Exclusion Criteria:

* Children afraid of clowns
* Children diagnosed with a mental, physical or visual impairment.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2017-04-30 (Estimated); Primary Completion 2017-06-30 (Estimated); Study Completion 2017-08-31 (Estimated)

PRIMARY OUTCOMES:
Acceptability | T3 (immediately after the procedure before leaving the treatment room)
  Acceptability will be assessed with parents and nurses using a satisfaction survey. The survey will be provided to parents in paper form and will be verbally completed by the nurse. In addition, to document the feasibility and acceptability of the study, the number of children participating, as well as the duration of the procedure and the number of professionals involved will be noted throughout the procedure.

SECONDARY OUTCOMES:
Pain intensity | T2 (during the immunization procedure)
  French version of the Face, Legs, Activity, Cry and Consolability (FLACC)
Anxiety Level | T1 (baseline), T2 (during the procedure).
  Visual Analogue Scale (VAS).

IPD SHARING:
Plan to Share IPD: No